CLINICAL TRIAL: NCT06617195
Title: Mechanisms of Anabolic Resistance in Older Humans
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian R. Lanza, Principal Investigator, Mayo Clinic
Other Study IDs: 24-003329
Record Dates: First submitted 2024-09-13; First posted 2024-09-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma Serum Adipose tissue Skeletal muscle tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: Men and women between the ages of 21-35 years will be recruited for this study. All participants will complete an outpatient study day (body composition, blood draw, treadmill test, strength test) and an inpatient study day (muscle biopsies, fat biopsies, indirect calorimetry, exercise test).
  Interventions: Other: Exercise
- Older: Men and women between the ages of 70-85 years will be recruited for this study. All participants will complete an outpatient study day (body composition, blood draw, treadmill test, strength test) and an inpatient study day (muscle biopsies, fat biopsies, indirect calorimetry, exercise test).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Young and older adults will perform a single bout of unaccustomed resistance exercise to evaluate molecular and cellular response in skeletal muscle

SUMMARY:
The purpose of this research is to understand how chronic inflammation affects muscle function and responses to exercise in older adults.

DETAILED DESCRIPTION:
Inflamed adipose tissue may contribute to blunted exercise response in skeletal muscle of older adults. The objective of this project is to evaluate a hypothesis that inflamed adipose secretes factors that activate inflammatory cascades in skeletal muscle, which may interfere with exercise-responsive molecular pathways and contribute to dysfunctional muscle phenotypes with aging. This project determine how adipose tissue influences skeletal muscle function and anabolic response to exercise in older adults. Young and older adults will complete studies to assess molecular response to acute exercise from protein synthesis rates, mRNA of exercise-responsive genes, and activation of signaling proteins in skeletal muscle. Adipose tissue will be assessed using a combination of non-invasive imaging and biopsy-based molecular phenotyping. The project will determine if acute exercise response is attenuated in older adults with inflamed adipose tissue phenotype.

ELIGIBILITY:
Exclusion Criteria:

1. Diabetes or fasting plasma glucose 126 mg/dL
2. Body mass index (BMI) 30 kg/m2
3. Anemia (female subjects hemoglobin of <11 g/dl and male subjects hemoglobin <12 g/dl)
4. Active coronary artery disease or history of unstable macrovascular disease (unstable angina, myocardial infarction, stroke, and revascularization of coronary, peripheral or carotid artery within 3 months of recruitment)
5. Renal failure (serum creatinine > 1.5mg/dl)
6. Chronic active liver disease (AST>144IU/L or ALT>165IU/L)
7. Oral warfarin group medications or history of blood clotting disorders.
8. Smoking
9. Pregnancy or breastfeeding
10. Alcohol consumption greater than 2 glasses/day or other substance abuse
11. Untreated or uncontrolled hypothyroidism
12. Debilitating chronic disease (at the discretion of the investigators)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women age 21-35 years or 70-85 years of age
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-09-16 (Estimated); Study Completion 2030-09-16 (Estimated)

PRIMARY OUTCOMES:
Anabolic response | 2 months
  Skeletal muscle protein synthesis rates will be measured from isotopic enrichment of muscle proteins

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lanza, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Anthropometric data Primary and secondary outcomes